CLINICAL TRIAL: NCT05806489
Title: Effect of Intermittent Fasting on Glycaemic Variability in Healthy Subjects
Brief Title: Glycemic Variability in Intermittent Fasting
Acronym: GLUInterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Banjari, Associate Professor, Clinical Nutrition Specialist, Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IBanjari-1
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Intermittent Fasting
Keywords: Blood Glucose; Glycemic variability; Intermittent fasting; Crossover Intervention
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting (Experimental)
  Interventions: Other: Intermittent Fasting
- Control Diet (Placebo Comparator)
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: Intermittent Fasting — Participants received a 3-day individualized diet plan consisting of 3 meals per day. Meals needed to be consumed during 6 hours (while fasting for the remaining 18 hours). Diet plans were matched for energy and macronutrients.
  Arms: Intermittent Fasting
Other: Control Diet — Participants received a 3-day individualized diet plan consisting of 3 meals per day. Meals needed to be consumed during 12 hours (while fasting for the remaining 12 hours). Diet plans were matched for energy and macronutrients.
  Arms: Control Diet

SUMMARY:
The aim was to test the difference in glycemic variability after meal consumption during intermittent fasting and the usual diet.

DETAILED DESCRIPTION:
Healthy participants were recruited for this crossover study aiming to determine the difference in glycemic variability after meal consumption while practicing intermittent fasting and the usual diet. Prior to the protocol assignment, participants were followed for 3 days - they were instructed to maintain their usual sleep pattern, level of physical activity and diet. Control of dietary pattern was conducted by using the 3-day food diary. Day zero was preparation day for the protocol (Intermittent fasting or Control diet) when all participants received individualized 3-day diet plan. Each protocol lasted 3 days with a 7-day washout period. Each protocol consisted of 3 meals per day, each providing a third of the total energy requirement. Control diet protocol was set at 12 hours eating/12 hours fasting, and Intermittent fasting protocol 6 hours eating/18 hours fasting. Blood glucose was measured at zero, 15, 30, 45 and 90 minutes after meal consumption. Before breakfast, blood glucose was measured also at minus 5 minutes prior meal consumption.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index in the range between 18.5 and 29.9 kg/m^2
* stable sleep pattern (going to bed between 21:30h and midnight)
* for women: regular menstrual cycle lasting between 21 and 35 days, with average bleeding time 2 to 6 days

Exclusion Criteria:

* Body Mass Index below 18.5 or above 29.9 kg/m^2
* irregular sleeping pattern
* work in nightshift
* high intensity workout routine
* irregular dietary patterns (e.g. skipping meals)
* regularly fasting for more than 15 hours per day
* diagnosis of diabetes (or other conditions related to glycemic disorders)
* hypertension or other cardiovascular disease
* neurologic conditions
* disease affecting metabolism (like liver, kidney, thyroid or lung)
* use of medications for glycemia, hypertension, steroids, adrenergic stimulators, laxatives or supplements affecting glycemia, circadian rhythm, sleep or metabolism in general

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 3 days per protocol
  Change in blood glucose
Glycemic variability | 3 days per protocol
  Coefficient of Variation expressed as the ratio between standard deviation and mean blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Ines Banjari, PhD, Principal Investigator — University of Osijek, Croatia
Locations (1):
- Department of Food and Nutrition Research, Faculty of Food Technology, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No
All the results will be published (as journal manuscript) and freely accessible to all interested parties. Also, interested parties can contact investigators for any details regarding the study and results (for example if individual data is required for a meta-analysis).